CLINICAL TRIAL: NCT07052279
Title: Water Based Burpee Exercises on Functional Capacity in Poste-menopausal Women After Thyroidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Mohamed Saied Zidan, Assistant professor doctor, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 2/4/2024-2025
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Burpee Exercise; Water Exercises; Functional Capacity; Postmenopausal; Thyroidectomy
Keywords: burpee exercises; postmenopausal; thyroidectomy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Control group will perform traditional aerobic exercises
  Interventions: Other: aerobic exercises
- Experimental group (Experimental): Experimental group will perform water based burpee exercises
  Interventions: Other: water based burpee exercises

INTERVENTIONS:
Other: water based burpee exercises — water based burpee exercises ( Aquatic exercise ) is one method that has previously been shown to improve muscle strength, balance, and coordination in those of advancing age Although the evidence supports the effectiveness of both water-based burpee exercise in middle-aged and elderly individuals, has, to our knowledge, never been investigated. Thus, the objective of this study was to assess the long-term effect of water-based burpee exercises
  Arms: Experimental group
Other: aerobic exercises — Traditional aerobic exercises for post-menopause include activities like brisk walking, jogging and cycling. These exercises help improve cardiovascular health, boost metabolism, and enhance mood. They can also be beneficial for maintaining bone density, especially weight-bearing exercises like walking and jogging.
  Arms: Control group

SUMMARY:
Skeletal muscle mass plays an important role with both metabolism and functional capacity. It is well established that the aging process leads to a significant decline in both muscle mass and strength which is associated with frailty , an increased risk of falls and decreased physical fitness and function In this context, high-load resistance training has been shown to reduce the risk of falls and increase strength and functional capacity in middle-aged and/or elderly individuals.

Aquatic exercise is one method that has previously been shown to improve muscle strength, balance, and coordination in those of advancing age Although the evidence supports the effectiveness of both water-based burpee exercise in middle-aged and elderly individuals, has, to our knowledge, never been investigated. Thus, the objective of this study was to assess the long-term effect of water-based burpee exercises

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 54 ± 4 years .

  * Post-menopausal women after tyhroidectomy
  * Body mass index (BMI) ≥ 30 kg/m².
  * Absence of osteoarticular dysfunctions in the lower limbs.
  * No personal history of cardiovascular disease
  * No water trauma
  * Non-smokers

Exclusion Criteria:

* History of Cardiovascular disorders.

  * Severe osteoarticular dysfunctions.
  * Presence of Water panic.
  * Participation in another clinical trial within the last 30 days.
  * Neurologic and psychiatric disorders (spina bifida, cerebral palsy, anorexia nervosa, known autism spectrum disorders).

Ages: 50 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC ( % ) | pre and post 8 weeks
  Description: The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. That can reflect pulmonary function , using portable spirometer ( SP 80B,China)
FEV1 ( liters ) | pre and post 8 weeks
  Forced expiratory volume in 1 second that can reflect pulmonary function , using portable spirometer ( SP 80B,China)
PEF ( liters / minute ) | pre and post 8 weeks
  Peak expiratory flow (PEF), a key indicator of lung function,using portable spirometer ( SP 80B,China)
FVC ( liters ) | Pre and post 8 weeks
  Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test. Forced expiratory volume and forced vital capacity are lung function tests , using portable spirometer ( SP 80B , China )
Chest expansion ( centimeter ) | Pre and post 8 weeks
  A simple, noninvasive pulmonary function test used to assess chest wall mobility and, to a lesser extent, lung function , using tape measurement.

SECONDARY OUTCOMES:
Timed up and go test ( seconds ) | Pre and post 8 weeks
  A simple, quick, and widely used clinical performance-based measure of functional mobility and fall risk. It assesses how long it takes for a person to rise from a chair, walk three meters, turn, walk back, and sit down again.
Gait Speed ( meters per second ) ( 4 Metre Walk Test ) | Pre and post 8 weeks
  Is the rate at which a person walks, is typically measured in meters per second (m/s). This is determined by dividing the distance walked by the time it takes to walk that distance. such as ( 4 Metre Walk Test )
30-Second Chair Test ( number of times the patient comes to a full standing position in 30 seconds ). | Pre and post 8 weeks
  Designed for testing leg strength and endurance in older adults.
Berg Balance Scale (BBS) to test dynamic balance | Pre and post 8 weeks
  A widely used assessment tool in physical therapy to evaluate a patient's functional balance and fall risk. It consists of 14 tasks, scored on a 5-point scale from 0 to 4, with a total possible score of 56. A lower score indicates a higher risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Saied Zidan, Cairo, Egypt